CLINICAL TRIAL: NCT04992273
Title: A Phase 2A, Open-Label Study Assessing Pharmacokinetics, Safety, Tolerability, and Immunogenicity of Single-Dose Subcutaneous Anti- Spike(s) SARS-COV-2 Monoclonal Antibodies (Casirivimab and Imdevimab) in High-Risk Pediatric Subjects Under 12 Years of Age
Brief Title: COVID-19 Administration of Single-Dose Subcutaneous Anti- Spike(s) SARS-CoV-2 Monoclonal Antibodies Casirivimab and Imdevimab in High-Risk Pediatric Participants Under 12 Years of Age
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Emerging SARS-CoV-2 variants impacting susceptibility to study drug
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R10933-10987-COV-2121; 2021-004590-30 (EudraCT Number); NCT05149300 (obsolete NCT alias)
Record Dates: First submitted 2021-08-03; First posted 2021-08-05 (Actual); Results first posted 2023-03-06 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: COVID-19
Keywords: Coronavirus disease 2019 (COVID-19); Severe acute respiratory syndrome coronavirus 2 (SARS-COV-2); coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — casirivimab and imdevimab drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ≥20 kg to <40 kg (Experimental): SC administration
  Interventions: Drug: casirivimab+imdevimab
- ≥10 kg to <20 kg (Experimental): SC administration
  Interventions: Drug: casirivimab+imdevimab
- ≥5 kg to <10 kg (Experimental): SC administration
  Interventions: Drug: casirivimab+imdevimab
- ≥3 kg to <5 kg (Experimental): SC administration
  Interventions: Drug: casirivimab+imdevimab

INTERVENTIONS:
Drug: casirivimab+imdevimab — Single dose administered based on weight
  Other Names: REGN10933-10987; REGN-COV2; REGEN-COV™; RONAPREVE™

SUMMARY:
The primary objective of the study is to characterize the concentrations of casirivimab+imdevimab in serum over time after a single subcutaneous (SC) administration

The secondary objectives of the study are:

* To assess the safety and tolerability of SC or single administration of casirivimab+imdevimab
* To assess the occurrence of grade ≥3 injection site reactions and grade ≥3 hypersensitivity reactions, in participants treated with SC doses of casirivimab+imdevimab
* To assess the immunogenicity of casirivimab+imdevimab

ELIGIBILITY:
Key Inclusion Criteria:

1. Is <12 years of age and ≥3 kg to <40 kg at the time parental/guardian consent is signed
2. Has at least one risk factor for developing severe COVID-19 if they were to become infected, such as:

   1. Obesity (BMI [kg/m2] ≥95th percentile for age and sex based on CDC growth charts)
   2. Cardiovascular disease
   3. Chronic lung disease
   4. Type 1 or type 2 diabetes mellitus
   5. Chronic kidney disease, including those on dialysis
   6. Chronic liver disease
   7. Immunocompromised or immunodeficient, based on Investigator's assessment (examples include cancer treatment, bone marrow or organ transplantation, immune deficiencies, HIV infection, sickle cell anemia, thalassemia, and prolonged use of immune-weakening medications)
   8. Medical complexities (examples include any underlying genetic condition, neurologic condition, metabolic condition, or congenital heart disease)
   9. Any other condition deemed by the Investigator to be a risk factor for severe COVID-19

Key Exclusion Criteria:

1. Has positive diagnostic test for SARS-CoV-2 infection from a sample collected during screening ≤7 days prior to study drug administration Note: The sample for the test should be collected ≤7 days within study drug administration, and the result should be reviewed and confirmed negative prior to dosing. Historical records will not be accepted.
2. Has active respiratory or non-respiratory symptoms consistent with COVID-19 in the opinion of the Investigator
3. Has subject-reported clinical history of COVID-19, as determined by Investigator, within the last 90 days
4. Has subject-reported history of prior Emergency Use Authorization (EUA)/approved positive diagnostic test for SARSCoV-2 infection within the last 90 days
5. Is currently hospitalized or was hospitalized for >24 hours for any reason within 14 days of the screening visit
6. Prior use (within 90 days prior to study drug administration) or current use of any investigational, authorized, or approved passive antibody for prophylaxis of SARS-CoV-2 infection, including convalescent plasma, convalescent sera, hyperimmune globulin, or other monoclonal antibodies (eg, bamlanivimab and etesevimab, sotrovimab)
7. Has initiated vaccination for SARS-CoV-2 with an investigational or approved vaccine, but has not completed the vaccine schedule as recommended by the vaccine manufacturer.
8. Plans to receive an investigational or approved SARS-CoV-2 vaccine within 90 days after study drug administration, or per the recommended time frame from the current Centers for Disease Control vaccination guidelines (CDC, 2021b)

NOTE: Other protocol-defined Inclusion/ Exclusion Criteria apply

Ages: 1 Minute to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (7):
- United States (7):
  - Advanced Research Center, Inc, Anaheim, California
  - Batchelor's Children's Research Institute, Miami, Florida
  - Stony Brook University Hospital, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Jacobi Medical Center, The Bronx, New York
  - Coastal Pediatric Research, Charleston, South Carolina
  - Regeneron Research Site, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 7 participants were screened. All 7 enrolled into Group A (≥10 kg to <40 kg). One discontinued at week 9 due to being lost to follow-up. Participants in Group A (≥10 kg to <40 kg) were subsequently divided into 2 groups for analysis: Group A1 (≥20 kg to <40 kg) and Group A2 (≥10 kg to <20 kg) and received different doses. Two participants enrolled in Group A1, 5 enrolled in Group A2; all 7 participants were enrolled and treated.
Groups:
- ≥20 kg to <40 kg; ≥10 kg to <20 kg: Single dose of casirivimab+imdevimab, that was the body weight dose equivalent to the 1200 mg adult dose (600 mg of casirivimab and 600 mg of imdevimab) administered as 1 to 4 subcutaneous (SC) injections based on body weight.
Period: Overall Study
Arm/Group | ≥20 kg to <40 kg | ≥10 kg to <20 kg
Started | 2 | 5
Completed | 2 | 4
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ≥20 kg to <40 kg | ≥10 kg to <20 kg | Total
Number analyzed (Participants) | 2 | 5 | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.5 (2.12) | 3.0 (1.58) | 4.9 (3.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 5 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 4 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of Casirivimab+Imdevimab in Serum Over Time.
Description: Concentrations reported in milligrams per Liter (mg/L)
Time Frame: Day 0 and Day 14
Population: Here 'n' = the number of evaluable participants at the specified time point
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- ≥10 kg to <40 kg: Single dose of casirivimab+imdevimab, that was the body weight dose equivalent to the 1200 mg adult dose administered as 1 to 4 subcutaneous (SC) injections based on body weight.
Arm/Group | ≥10 kg to <40 kg
Number analyzed (Participants) | 7
mg/L
  Day 0 | 0 (0)
  Day 14 | 239.0 (36.3)

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Time Frame: Through end of study, approximately 24 weeks
Population: The Safety Analysis Set (SAF) includes all participants who received any study drug; it is based on the treatment received (as treated).
Measure: Count of Participants; unit: Participants
Arm/Group | ≥20 kg to <40 kg | ≥10 kg to <20 kg
Number analyzed (Participants) | 2 | 5
Participants | 2 | 3

3. Secondary Outcome: Number of Participants With Indicated Severity of TEAEs
Description: Treatment-emergent adverse events (TEAEs) are defined as those that are not present at baseline or represent the exacerbation of a pre-existing condition during the on-treatment period. The severity of AEs were graded using version 5.0 of NCI-CTCAE.
Time Frame: Through end of study, approximately 24 weeks
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | ≥20 kg to <40 kg | ≥10 kg to <20 kg
Number analyzed (Participants) | 2 | 5
Participants
  Infections and Infestations - Grade 1 | 1 | 1
  Infections and Infestations - Grade 2 | 1 | 1
  Infections and Infestations - Grade 3 | 0 | 0
  Infections and Infestations - Grade 4 | 0 | 0
  Infections and Infestations - Grade 5 | 0 | 0
  Respiratory, thoracic and mediastinal disorders - Grade 1 | 0 | 1
  Respiratory, thoracic and mediastinal disorders - Grade 2 | 1 | 1
  Respiratory, thoracic and mediastinal disorders - Grade 3 | 0 | 0
  Respiratory, thoracic and mediastinal disorders - Grade 4 | 0 | 0
  Respiratory, thoracic and mediastinal disorders - Grade 5 | 0 | 0
  Nervous system disorders - Grade 1 | 0 | 1
  Nervous system disorders - Grade 2 | 0 | 0
  Nervous system disorders - Grade 3 | 0 | 0
  Nervous system disorders - Grade 4 | 0 | 0
  Nervous system disorders - Grade 5 | 0 | 0

4. Secondary Outcome: Number of Participants With Grade ≥3 Injection Site Reactions
Time Frame: Through Day 4
Measure: Count of Participants; unit: Participants
Arm/Group | ≥20 kg to <40 kg | ≥10 kg to <20 kg
Number analyzed (Participants) | 2 | 5
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With Grade ≥3 Hypersensitivity Reactions
Time Frame: Through Day 4
Measure: Count of Participants; unit: Participants
Arm/Group | ≥20 kg to <40 kg | ≥10 kg to <20 kg
Number analyzed (Participants) | 2 | 5
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Indicated Immunogenicity as Measured by Anti-drug Antibodies (ADA) to Casirivimab Over Time
Time Frame: Up to 24 weeks
Population: Here 'n' = number of evaluable participants at the specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | ≥20 kg to <40 kg | ≥10 kg to <20 kg
Number analyzed (Participants) | 2 | 4
Participants | 2 | 3

7. Secondary Outcome: Number of Participants With Indicated Immunogenicity as Measured by ADA to Imdevimab Over Time
Time Frame: Up to 24 weeks
Population: Here 'n' = number of evaluable participants at the specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | ≥20 kg to <40 kg | ≥10 kg to <20 kg
Number analyzed (Participants) | 2 | 4
Participants | 2 | 3

8. Secondary Outcome: Immunogenicity as Measured by Neutralizing Antibodies (NAb) to Casirivimab Over Time
Time Frame: Up to 24 weeks
Population: Neutralizing antibody (NAb) analysis data was not collected.
Arm/Group | ≥20 kg to <40 kg | ≥10 kg to <20 kg
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Immunogenicity as Measured by NAb to Imdevimab Over Time
Time Frame: Up to 24 weeks
Population: Neutralizing antibody (NAb) analysis data was not collected.
Arm/Group | ≥20 kg to <40 kg | ≥10 kg to <20 kg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose to week 24
Groups:
- Group A1 ≥ 20 kg to <40 kg; Group A2 ≥ 10 kg to <20 kg: Single dose of casirivimab+imdevimab, that was the body weight dose equivalent to the 1200 mg adult dose (600 mg of casirivimab and 600 mg of imdevimab) administered as 1 to 4 subcutaneous (SC) injections based on body weight.
Arm/Group | Group A1 ≥ 20 kg to <40 kg | Group A2 ≥ 10 kg to <20 kg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/5
Other Adverse Events (participants affected / at risk) | 2/2 | 3/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A1 ≥ 20 kg to <40 kg (N=2) | Group A2 ≥ 10 kg to <20 kg (N=5)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough variant asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
The study was terminated early due to emerging SARS-CoV-2 variants impacting susceptibility to the study drug. The early termination was not due to safety findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT04992273/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT04992273/SAP_001.pdf